CLINICAL TRIAL: NCT07278921
Title: Retrospective, Multicenter Observational Study to Evaluate the Response to Treatment With Mosunetuzumab in Relapsed/Refractory Follicular Lymphoma (FL) After at Least Two Lines of Therapy, Within the Compassionate Use Program (CUP).
Brief Title: Study to Evaluate the Response to Treatment With Mosunetuzumab in Relapsed/Refractory Follicular Lymphoma (FL) After at Least Two Lines of Therapy, Within the Compassionate Use Program (CUP).
Acronym: MosuOSSHSR
Status: Recruiting | Type: Observational
Sponsor: Andrés José Maria Ferreri (Other)
Responsible Party: Sponsor-Investigator, Andrés José Maria Ferreri, Prof., IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: MosuOSSHSR
Record Dates: First submitted 2025-11-21; First posted 2025-12-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Mosunetuzumab — Adult patients (>18 years) with Follicular Non-Hodgkin Lymphoma, who have undergone at least two lines of therapy, treated with Mosunetuzumab under a compassionate use program

SUMMARY:
Retrospective, multicenter observational study to evaluate the response to treatment with Mosunetuzumab in relapsed/refractory Follicular Lymphoma (FL) after at least three lines of therapy, within the Compassionate Use Program (CUP).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) with follicular non-Hodgkin's lymphoma, undergoing at least two lines of therapy, treated with mosunetuzumab under a compassionate use program.
* Patients who have signed informed consent for treatment.

Exclusion Criteria:

* Age <18 years
* Patients with other types of cancer/lymphoma
* Patients not eligible for the Mosunetuzumab compassionate use program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Descriptive study of the Italian experience with the compassionate use of mosunetuzumab.
  Sample size: approximately 25 patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the response to Mosu (Lugano criteria) | Up to 1 year from treatment initiation
  The primary objective of the study is to evaluate the response to mosunetuzumab in patients diagnosed with follicular lymphoma from second-line therapy, within the national compassionate use program (CUP). This response is assessed according to the 2014 Lugano criteria.
Disease-free survival (PFS) | 1 year after starting treatment (PFS at 1 year)
  Disease-free survival (PFS) at 1 year is evaluated.

SECONDARY OUTCOMES:
OS | 12 month
  The study's secondary objective is to evaluate the overall survival (OS) of the included patients.
rate of toxicity | 12 months
  Analyze the rate of toxicity recorded during therapy, with particular attention to infusion reactions, CRS, and ICANS.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No